CLINICAL TRIAL: NCT06025552
Title: A First-in-Human (FIH), Randomized, Double-Blind, Placebo-controlled, Phase 1a Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Activity of TU7710 Following Single, Ascending, Intravenous, Dose Administration in Warfarin Anti-coagulated Healthy Male Subjects
Brief Title: Study of TU7710 in Warfarin Anti-coagulated Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TiumBio Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: TUB4PI-01
Record Dates: First submitted 2023-07-31; First posted 2023-09-06 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Hemophilia a; Hemophilia B; Blood Coagulation Disorders
MeSH Terms: conditions — Hemophilia A; Hemophilia B; Blood Coagulation Disorders | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: 5 cohorts with 5 dose levels will sequentially be escalated after safety review.
  8 subjects in each cohort who will be randomly assigned to placebo or TU7710 group in 2:6 ratio.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TU7710 (Experimental): TU7710 of escalating 5 doses
  Interventions: Drug: TU7710
- Normal Saline (placebo of TU7710) (Placebo Comparator): Placebo of TU7710 at corresponding TU7710 dose level
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: TU7710 — In each dose level, 6 subjects will be assigned to TU7710. Anticipated escalating dose levels are 100mcg/kg, 200mcg/kg, 400mcg/kg, 800mcg/kg and the last dose will be decided after assessing cohort 1~4 PK, PD, safety, and exploratory efficacy data.
  Arms: TU7710
Drug: Normal saline — Placebo of TU7710 at corresponding TU7710 dose level. In each dose level, 2 subjects will be assigned to placebo group.
  Arms: Normal Saline (placebo of TU7710)

SUMMARY:
This is a Phase 1a, double-blind, randomized, placebo- controlled, SAD study to assess safety, tolerability, PK, and PD of TU7710 in warfarin treated healthy male participants.

DETAILED DESCRIPTION:
The 40 subjects will be divided into 5 cohorts, and the subjects assigned to each cohort will be randomly assigned with 6 persons receiving TU7710 and 2 persons receiving a placebo for TU7710. Each cohort will proceed in sequence and the next cohort study will be decided by the Safety Monitoring Committee (SMC) .

Subjects will be participated in the study after warfarin anti-coagulation to maintain the INR between 2.00 and 3.00 as a preventive measure for potential thrombosis prior to the IP administration.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥19 and ≤45
* BMI of ≥18.0 kg/m2 and ≤30.0 kg/m2
* Body weight of ≥55.0 kg and ≤90.0 kg
* Provide informed consent and willing to comply with study requirements.

Exclusion Criteria:

* History or at risk of developing diseases related to venous thromboembolic events or has family history of such disease
* History of major bleeding/traumatic event or major surgery within 6 month
* History of any other clinically relevant coagulation disorder (such as gastrointestinal bleeding, hemorrhoid hemorrhage)
* Abnormal coagulation related laboratory abnormal test results, including protein C, protein S, PT, aPTT
* history or current symptoms of gastrointestinal, liver, or renal disease that may affect the pharmacokinetics of the IP
* History of or are currently with hepatitis B or C (active or carrier state) or human immunodeficiency virus (HIV) or syphilis infection.
* Currently smoking or have smoked within 1 month before IP or positive cotinine results
* History of alcohol abuse or positive alcohol breath test
* Excessive caffeine intake within 7 days before IP
* INR results not between 2.0~3.0 range after warfarin treatment
* History of hypersensitivity to medicinal product similar to TU7710 active ingredient or excipient
* Laboratory abnormal test results, such as QTcF <340msec or >450msec (or family history of long QT syndrome), LDL >190mg/dl , Total cholesterol >300mg/dl, triglycerides > 350mg/dl, ALT >1.5*ULN, AST >1.5*ULN, bilirubin >1.5*ULN
* Abnormal vital sign SBP >140mmHG, DBP <90mmHg, heart rate <40bpm or >85bpm
* Any medical history that may increase the risk or affect the evaluation of study objectives by participating in this study at the discretion of the investigator. (e.g., neurology or psychiatric history)

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
Number and proportion of participants with adverse events | 30 days post-dose
  Number and proportion of participants with adverse events/ adverse reaction /SAE overall and by treatment group
Number of subjects with significant abnormal laboratory values | 30 days post-dose
  Mean with standard deviation, median, maximum, minimum results of laboratory values in each treatment group. The laboratory parameters that will be assessed are clinical chemistry, hematology and urinalysis.
ADA and Neutralizing antibody results | 30 days post-dose
  Incidence of subjects with ADA and Nab positive results
Number of subjects with significant abnormal Electrocardiography (ECG) findings | 30 days post-dose
  Mean with standard deviation, median, maximum, minimum results of ECG results in each treatment group. The ECG parameters that will be assessed are heart rate, PR interval, QRS interval, QT interval, and QTcF interval.
Number of subjects With Significant Abnormal vital sign findings | 30 days post-dose
  Mean with standard deviation, median, maximum, minimum results of vital sign values in each treatment group. The vital signs that will be assessed are body temperature, pulse rate, respiratory rate, and systolic and diastolic blood pressure.

SECONDARY OUTCOMES:
Pharmacokinetics assessment_Maximum concentration | 4 days post-dose
  Maximum plasma VIIa activity level in each dose level
Pharmacokinetics assessment_AUC last | 4 days post-dose
  Area under plasma activity-time curve after TU7710 single administration from time zero to last quantifiable concentration
Pharmacokinetics assessment_AUC inf | 4 days post-dose
  Area Under the Plasma activity-time curve after TU7710 single administration From Time Zero Extrapolated to Infinity
Pharmacokinetics assessment_Clearance | 4 days post-dose
  Clearance after TU7710 single administration
Pharmacokinetics assessment_Volume of distribution | 4 days post-dose
  Volume of distribution after TU7710 single administration
Pharmacokinetics assessment_Dose proportionality | 4 days post-dose
  Regression analysis using the power model between the log-converted Cmax, AUClast, and the log-converted dose can be performed, and each parameter adjusted by dose can be calculated and compared between the dose groups
Pharmacokinetics assessment_Tmax | 4 days post-dose
  Time from administration to maximum plasma VIIa level in each dose level
Pharmacodynamic assessment_INR change from baseline | 5 days post-dose
  INR measurement change from baseline to day 5 in each treatment group and dose level
Pharmacodynamic assessment_PT change from baseline | 5 days post-dose
  PT measurement change from baseline to day 5 in each treatment group and dose level
Pharmacodynamic assessment_aPTT change from baseline | 5 days post-dose
  aPTT measurement change from baseline to day 5 in each treatment group and dose level
Pharmacokinetics assessment_incremental recovery | 4 days post-dose
  Incremental recovery after TU7710 single administration expressed as the ratio of measured peak level against dose per bodyweight

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea